CLINICAL TRIAL: NCT02297217
Title: A Phase 2 Study of Palliative Chemo-Radiotherapy With Carbo-Taxol in Non-Curative Cancer of the Esophagus
Brief Title: Chemoradiotherapy for Advanced Esophageal Cancer
Acronym: PaRCUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Principal Investigator, Marc Kerba, MD, AHS Cancer Control Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CC-14-0122
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy with Concurrent Radiation (Experimental): Carboplatin and paclitaxel will be administered intravenously on Days 1 and 8 while radiation therapy is administered
  Interventions: Drug: Carboplatin and Taxol (paclitaxel); Radiation: External Beam Radiation

INTERVENTIONS:
Drug: Carboplatin and Taxol (paclitaxel) — Patients will receive carboplatin (AUC 2) and paclitaxel (50 mg/m2) intravenously on Days 1 and 8. Patients are seen for 2 weekly Treatment Visits during concurrent chemo-radiation then every 28 days until the End of Study Visit, approximately 6 months after Treatment Visit 1. Preparation and administration of chemotherapy will be according to local site standard of care.
Radiation: External Beam Radiation — Patients will receive external beam radiation therapy of 30Gy/10 fractions over two weeks (or reduced to 25 Gy/10 fractions if acute toxicity parameters are met during the run-in) and receive carboplatin (AUC 2) and paclitaxel (50 mg/m2) intravenously on Days 1 and 8. Treatment will be planned, prescribed and delivered using standard 3D radiotherapy planning techniques to encompass the primary tumor and surrounding clinical target volume. Patients are seen for 2 weekly Treatment Visits during concurrent chemo-radiation then every 28 days until the End of Study Visit, approximately 6 months after Treatment Visit 1.

SUMMARY:
This study aims to show that the addition of carboplatin and paclitaxel chemotherapy to a palliative course of external beam radiation treatment improves both dysphagia relief and patient quality of life in patients with unresectable esophageal cancer.

DETAILED DESCRIPTION:
Patients with carcinoma of the esophagus not suitable for definitive radical treatment who have symptomatic dysphagia requiring locoregional palliation, and who have no contra-indications to chemo-radiotherapy will be offered Carboplatin (AUC 2) and paclitaxel (50 mg/m2) intravenously on days 1 and 8 concurrent with external beam radiation therapy of 30Gy/10 fractions over two weeks where the primary goal is relief of dysphagia and other outcomes include toxicity, quality of life and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven carcinoma of the esophagus.
2. Not a candidate for radical/curative treatment due to the advanced nature of the disease, presence of metastases, or intercurrent illness.
3. Symptomatic patients with Mellow Dysphagia Scores of ≥ 1 i.e. able to eat only some solids.
4. ECOG Performance status ≤ 2.
5. Patients able to begin treatment within 14 days of signing the informed consent form.
6. Patient is at least 18 years old.
7. Hematological function as defined by the following laboratory parameters:

   * Hemoglobin > 100g/L
   * Platelet count > 100x10E9/L
   * Absolute neutrophil count > 1.5x10E9/L
8. Renal function to undergo chemotherapy as defined by the following laboratory parameters:

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x the upper limit of institutional normal (≤ 5 if liver metastases)
   * Total bilirubin ≤ 1.5x the upper limit of institutional normal
   * Calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault formula
9. Patients capable of childbearing are using adequate contraception.
10. Written and informed consent of patient.

Exclusion Criteria:

1. Previous radiotherapy delivered to the chest.
2. Synchronous active malignancies.
3. Pregnant or lactating patients: women of child bearing potential must have a negative serum pregnancy test within 7 days of Treatment Visit 1. Women or men of child bearing potential must use effective contraception (defined by the use of two birth control methods, which can be either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy). Subjects must start using birth control from the time they have signed the Informed Consent Form prior to start of therapy until 120 days post completion of study therapy or study discontinuation, which must be documented in the eCRF.
4. Patients unfit for any treatment component, including absolute contraindications for radiotherapy or Connective Tissue Disease.
5. Tracheo-esophageal fistula.
6. Esophageal stents in situ.
7. Previous chemotherapy for esophageal cancer
8. Unable to complete surveys in English without aid of interpreter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve relief of dysphagia | up to day 85
  Will be measured as the proportion of patients who achieve relief of dysphagia, defined as improvement of at least one point on the Mellow Dysphagia Score, measured at Day 57 after the start of radiotherapy, and maintained for at least 28 calendar days (until the Day 85 visit).

SECONDARY OUTCOMES:
Dysphagia progression free survival | 6 Months
  Will be measured from screening to the time of first progression of dysphagia. Progression of dysphagia will be defined as follows:
  * A drop of at least 1 point on the 5 point Mellow Dysphagia Score,
  * Stricture requiring intervention, or
  * Death,
  Other secondary objectives as follows:
  Time to achieving any response in dysphagia after treatment as measured by an improvement of at least 1 point on the 5 point Mellow Dysphagia Score. Number of patients receiving secondary treatment (radiation, chemotherapy or stenting), Utility assessments pre to post treatment and at 3 and 6 months, Quality of life differences post treatment and at 3 and 6 months. Measures of biological/serological correlates of response, Acute and late toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kerba, MD, Principal Investigator — 5872316617
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada